CLINICAL TRIAL: NCT03341026
Title: An Open, Multicenter, Randomized, Controlled Pilot Trial Evaluating the Metronom Continuous Glucose Monitoring System in Subjects With Type 1 Diabetes Mellitus
Brief Title: Metronom Continuous Glucose Monitoring System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Metronom Health (Industry)
Collaborators: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ELITE02
Record Dates: First submitted 2017-10-30; First posted 2017-11-14 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabete Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction day 1, 4, 7, 14 (Other): Patient will come to the hospital on day 1, 4, 7 and 14. A hypo- or hyperglycaemic experiment will start according to allocation by randomizer.
  Interventions: Other: Metronom CGM device
- Induction day 1, 7, 10, 14 (Other): Patient will come to the hospital on day 1, 7, 10 and 14. A hypo- or hyperglycaemic experiment will start according to allocation by randomizer.
  Interventions: Other: Metronom CGM device

INTERVENTIONS:
Other: Metronom CGM device — Patient receives three Metronom CGM devices on day 1. On day 1, 4, 7 and 14, a hypo- or hyperglycaemic experiment will start according to allocation by randomizer.
  Arms: Induction day 1, 4, 7, 14
Other: Metronom CGM device — Patient receives three Metronom CGM devices on day 1. On day 1, 7, 10 and 14, a hypo- or hyperglycaemic experiment will start according to allocation by randomizer.
  Arms: Induction day 1, 7, 10, 14

SUMMARY:
The aim of the present study is to investigate the clinical performance of the Metronom CGM system in patients with type 1 diabetes over a period of 14 days. In this study, the CGM sensor will be tested in an inpatient setting (meal/insulin test with frequent plasma glucose monitoring) at different days of wear-time. Sensor data will be compared to gold standard reference (Super GL2 analyser or YSI) and stability of sensor performance will be assessed over time. Additionally, safety and tolerability of the sensor will be investigated by regular assessment of the insertion site.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained after being advised of the nature of the study
* Male or female aged ≥18 years
* Type 1 diabetes for at least 6 months according to the WHO definition treated with multiple daily injections (MDI) or continuous subcutaneous insulin infusion (CSII) for at least 3 months (for T1D only)
* Body Mass Index (BMI) <35 kg/m²
* Flash or continuous glucose monitoring (FGM, CGM) user
* Willing and able to wear the Metronom CGM System for the duration of the study and undergo all study procedures
* HbA1c ≤86 mmol/mol

Exclusion Criteria:

* Any disease or condition which the investigator or treating physician feels would interfere with the trial or the safety of the subject
* Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods
* Any mental condition rendering the subject incapable of giving his consent
* Subject is using any medication that significantly impacts glucose metabolism (oral steroids) except if stable for at least the last three months and expected to remain stable for the study duration
* Has severe medical or psychological condition(s) or chronic conditions/infections that in the opinion of the Investigator would compromise the subject's safety or successful participation in the study
* Subject is actively enrolled in another clinical trial
* Known adrenal gland problem, pancreatic tumour, or insulinoma
* Known bleeding disorder
* Known hypersensitivity to adhesive or skin lesions that hinder sensor insertion
* Inability of the subject to comply with all study procedures
* Inability of the subject to understand the subject information
* Subject donated blood in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 14 days
  Overall percentage of sensor values which fall within ± 20 mg/dl of the mean reference values at glucose concentrations <100 mg/dl and within ± 20% at glucose concentrations
  ≥100 mg/dl

SECONDARY OUTCOMES:
Reliability | 14 days
  Percentage of sensor values which fall within ± 20 mg/dl of the mean reference values at glucose concentrations <100 mg/dl and within ± 20% at glucose concentrations
  ≥100 mg/dl on different days of wear-time
Reliability | 14 days
  Percentage of sensor values which fall within ± 15 mg/dl of the mean reference values
  ≥100 mg/dl (cf. ISO 15197: 2013, Chapter 6.3.3) (overall, on different days of wear-time)
Reliability | 14 days
  Percentage of sensor values which fall within ± 30 mg/dl of the mean reference values at glucose concentrations <100 mg/dl and within ± 30% at glucose concentrations
  ≥100 mg/dl (overall, on different days of wear-time)
Reliability | 14 days
  Percentage of sensor values which fall within ± 40 mg/dl of the mean reference values at glucose concentrations <100 mg/dl and within ± 40% at glucose concentrations
  ≥100 mg/dl (overall, on different days of wear-time)
Accuracy | 14 days
  Overall percentage of test-to-reference measurement pairs with an Absolute Relative Difference (ARD) ≤15%.
Reliability | 14 days
  Percentage of test-to-reference measurement pairs with an Absolute Relative Difference (ARD) ≤15% (overall, on different days of wear-time)
Reliability | 14 days
  Mean (MARD) and Median Absolute Relative Difference (MedARD) (overall, on different days of wear-time)
Reliability | 14 days
  Mean (MARD) and Median Absolute Relative Difference (MedARD) with regard to reference measurements in the hypoglycaemic (≤70mg/dl), euglycaemic (70- 180mg/dl), and hyperglycaemic (≥180mg/dl) area (overall, on different days of weartime)
Reliability | 14 days
  Bland-Altman analysis comparing sensor values with reference measurements (overall, on different days of wear-time)
Reliability | 14 days
  Distribution of data points in the Point and Rate Error Grid (overall, on different days of wear-time)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Mader, Ass Prof, Principal Investigator — Medical University of Graz
Locations (2):
- Medical University of Graz, Graz, Austria
- Steno diabetes center, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No